CLINICAL TRIAL: NCT03772067
Title: Influence of Dairy Protein Breakfast on Overall Daily Glycemia, Weight Loss HbA1c and Clock Genes mRNA Expression, in Type 2 Diabetes
Brief Title: Influence of Dairy Protein Breakfast on Glycemia, Weight Loss and Clock Genes in T2D
Acronym: Mdiet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Zohar Landau (Unknown); Shani Tsameret (Unknown)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0226-17-WOMC
Record Dates: First submitted 2018-12-08; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Type2 Diabetes; Healthy Obesity, Metabolically
MeSH Terms: conditions — Obesity, Metabolically Benign | interventions — Continuous Glucose Monitoring; Insulin Secretion; Weights and Measures

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBdiet (Experimental): This arm consist on 3 month on Bdiet with high energy and protein breakfast (660 +/-20 kcal), medium sized lunch (580+/-20 kcal) and dinner reduced in energy (300+/-20 kcal), with distribution of calories: breakfast 44%, lunch 37% and dinner 19%. The breakfast will contain 38 g protein mostly from milk and dairy products.
  Interventions: Device: Continuous glucose monitoring CGM; Diagnostic Test: Clock Genes m RNA expression; Diagnostic Test: Postprandial Glucose; Diagnostic Test: Postprandial Insulin; Diagnostic Test: Plasma GLP-1; Diagnostic Test: DPP4 plasma activity; Diagnostic Test: Ghrelin; Diagnostic Test: Plasma CCK; Diagnostic Test: Plasma PYY; Other: Body Weight; Diagnostic Test: Blood levels of HbA1c
- OBdiet (Active Comparator): This arm consist on 3 month on Bdiet with high energy and protein breakfast (660 +/-20 kcal), medium sized lunch (580+/-20 kcal) and dinner reduced in energy (300+/-20 kcal), with distribution of calories: breakfast 44%, lunch 37% and dinner 19%. The breakfast will 38 g protein without milk or dairy products mostly from other proteins, i.e. eggs, tuna, soy, oatmeal. Milk product will be avoided in this diet also in other meals along the day.
  Interventions: Device: Continuous glucose monitoring CGM; Diagnostic Test: Clock Genes m RNA expression; Diagnostic Test: Postprandial Glucose; Diagnostic Test: Postprandial Insulin; Diagnostic Test: Plasma GLP-1; Diagnostic Test: DPP4 plasma activity; Diagnostic Test: Ghrelin; Diagnostic Test: Plasma CCK; Diagnostic Test: Plasma PYY; Other: Body Weight; Diagnostic Test: Blood levels of HbA1c

INTERVENTIONS:
Device: Continuous glucose monitoring CGM — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the overall glucose levels measured with CGM installed in the arm during 14 days at baseline before diet intervention and after 14 days of the beginning of diet intervention
  Other Names: CGM
Diagnostic Test: Clock Genes m RNA expression — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the blood levels of Clock Genes measured at baseline and after 14 days of diet intervention
  Other Names: CG
Diagnostic Test: Postprandial Glucose — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial plasma Glucose measured at meal test after 14 days of diet intervention
  Other Names: PPG
Diagnostic Test: Postprandial Insulin — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial plasma Insulin measured at meal test after 14 days of diet intervention
  Other Names: Insulin
Diagnostic Test: Plasma GLP-1 — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial plasma GLP-1 measured at meal test after 14 days of diet intervention
  Other Names: GLP-1
Diagnostic Test: DPP4 plasma activity — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial DPP4 plasma activity measured at meal test after 14 days of diet intervention
  Other Names: DPP4
Diagnostic Test: Ghrelin — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial plasma Ghrelin measured at meal test after 14 days of diet intervention
Diagnostic Test: Plasma CCK — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial plasma CCK measured at meal test after 14 days of diet intervention
  Other Names: CCK
Diagnostic Test: Plasma PYY — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the postprandial plasma PYY measured at meal test after 14 days of diet intervention
  Other Names: PYY
Other: Body Weight — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing the body weight at baseline and every weeks of diet intervention
  Other Names: Weight
Diagnostic Test: Blood levels of HbA1c — The effect of the two diets (MBdiet and OBdiet) will be compared on the efficacy on changing blood HbA1c measured at baseline and after 90 days of diet intervention diet intervention
  Other Names: HbA1c

SUMMARY:
This study in T2D patients is undertaken to evaluate the effect of previously studied 3Meals Diet, high energy breakfast (Bdiet) with milk and dairy proteins (MBdiet) versus isocaloric diet with same meal distribution but with other sources of protein (OBdiet) overall postprandial glycemia (PPG), weight loss (WL), HbA1c, CG expression and on PPG, insulin, C-peptide, GLP-1, gut peptide YY (PYY), cholecystokinin (CCK), ghrelin, dipeptidyl peptidase-4 plasma activity (DPP-4) and appetite responses after high protein breakfast. challenge including milk and dairy products (MBdiet) and after breakfast challenge with same protein content but different source of protein (OBdiet)

DETAILED DESCRIPTION:
Increased circadian glucose excursions and overall postprandial glycemia (PPG) are linked to HbA1c and cardiovascular risk in T2D.

Most of the metabolic pathways involved in PPG i.e. secretion of insulin and glucagon-like peptide-1 (GLP-1), are controlled by circadian clock genes (CG). However, the CG regulation is bidirectional, indeed high protein breakfast (B), by increasing insulin and GLP-1 upregulate CG expression leading to reduced overall PPG, HbA1c and weight loss (WL) in T2D. Furthermore in recent study the investigators have shown that in type 2 diabetic patient treated with insulin a diet with 3 Meal Diet consisting in high energy and protein breakfast, medium sized lunch and low energy dinner, with selective time restriction from carbohydrate consumption after 15:00, designed as Bdiet; was more effective approach for reduction of overall PPG, HbA1c and for upregulation of Clock Genes (CG) mRNA expression compared to isocaloric 6 Meal Diet, with calories and macronutrient evenly distributed along the day in three main meals and 3 snack in between.

As the beneficial effects of high energy and protein breakfast in 3Meal diet on the reduction of body weight, overall glycemia and up regulation CG expression, have been demonstrated, in recent studies, we hypothesized that some sources of protein in the breakfast may exert be more beneficial than other source of protein on body weight, PPG, HbA1c and on CG expression Milk consumption is linked to lower risk for obesity and T2D. In acute studies, the addition of milk to carbohydrates in B, displayed greater lowering effect of glucose response after breakfast, lunch and dinner compared with other protein sources.

However the effect of a diet 3Mdiet with high energy and dairy protein breakfast (MBdiet), on overall PPG, weight loss HbA1c, the effect on effect on circadian clock genes and AMPK mRNA expression and on the postprandial glucose, insulin, C-peptide, GLP-1, PYY, CCK, ghrelin, DPP4 plasma activity and appetite has never been explored and never were compared to isocaloric 3Mdiet with other then dairy protein source of protein (OBdiet) in long term study in T2D individuals .

The investigators hypothesize that a diet with high energy and protein breakfast consisting on milk and dairy proteins (MBdiet), by enhancing clock gene expression will lead to more efficient weight loss reduction of overall PPG, and glucose control (HbA1c), compared to a diet with other (non dairy) proteins in the breakfast (OBdiet). The investigators also hypothesize that the dairy breakfast effects in MBdiet may be mediated, at least in part, by integration of events that promote greater postprandial glucose insulin, C-peptide, GLP-1, PYY, and CCK, and greater suppression of ghrelin appetite and DPP4 plasma activity,

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with T2D < 20 years;
* HgA1c ≥ 7.0 %.
* BMI - 28-40 kg/m2
* Men and women 30 -75 years of age inclusive.
* Normal liver, kidney and thyroid functions, negative urinary microalbumin test (urMA) and estimated glomerular filtration rate (eGFR) > 45 mL/min/1.73 m2.
* Type 2 diabetes controlled with diet and lifestyle alone or with antidiabetic treatment other than insulin (i.e. buguanides, sulfonylureas, glinides, SGLT2 inhibitors, DPP4 inhibitors, GLP-1 analogs), with stable doses for at least 3 months before entering the study.
* Stable weight (less than 5% change in body weight in last 3 months before the study - determined by self-reporting or documentation in clinical records).
* Concomitant medication i.e. antihypertensive, anti-lipidemic, anti-thrombotic drugs will be allowed also on stable dose for at least 3 months before the beginning of the trial.
* Patients that usually wake up between 06:00 and 08:00 and go to sleep between 22:00 and 24:00.
* Should not have shift work within 6 month of the study and should not have crossed time zones within 2 weeks of the study.

Exclusion Criteria:

* Type 1 diabetes or secondary forms of diabetes.
* Patients with latent autoimmune diabetes in adults (LADA).
* Treatment with insulin.
* Serum creatinine level >2mg/dl. Renal dysfunction: (estimated glomerular filtration rate eGFR < 45 mL/min/1.73 m2).
* Hepatic dysfunction: liver disease or transaminase levels > 2.5-fold above normal. Major illness with life expectancy < 5 years.
* Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer). Those taking psychotropic, anorectic medication, steroid treatment or with illicit drug abuse or alcoholism within one year prior to study onset. Pregnancy or lactation. Known hypersensitivity to milk components or lactose intolerance. Night or rotating shift workers or those who crossed more than 2 time zones during the 2- week period prior to study onset. No change in medication or nutrition supplements or physical activity will be made during the study. Not able to give informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-28 (Estimated); Primary Completion 2019-06-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Clock genes mRNA expression | two weeks
  The effect of the two diets (MBdiet and OBdiet) will be compared on their efficacy on changing the clock genes expression

SECONDARY OUTCOMES:
Continuous Glucose Monitoring (CGM) | two weeks
  The effect of the two diets (MBdiet and OBdiet) will be compared on their efficacy on changing overall glycemia assessed by Continuous Glucose Monitoring (CGM)
HbA1c | 3 months
  The effect of the two diets (MBdiet and OBdiet) will be compared on their efficacy on changing HbA1c
Body Weight | 3 months
  The effect of the two diets (MBdiet and OBdiet) will be compared on their efficacy on changing body weight

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Diabetes Unit E. Wolfson Hospital, Holon, Tel Aviv
  - Daniela Jakubowicz, Holon, Wolfson Medical Center

REFERENCES:
- [Derived] Tsameret S, Froy O, Matz Y, Landau Z, Twito O, Wainstein J, Avital-Cohen N, Chapnik N, Jakubowicz D. Glycaemic, appetite and circadian benefits of a dairy-enriched diet with high-protein breakfast and early daytime-restricted carbohydrate intake in type 2 diabetes: a randomised crossover trial. Diabetologia. 2026 Jan 23. doi: 10.1007/s00125-025-06658-2. Online ahead of print. PMID 41578008